CLINICAL TRIAL: NCT06119347
Title: Acute Kidney Injury in Cancer Patients Receiving Anti-Vascular Endothelial Growth Factor Monoclonal Antibody vs Immune Checkpoint Inhibitors: a Retrospective Real-world Study
Brief Title: Acute Kidney Injury in Cancer Patients Receiving Anti-Vascular Endothelial Growth Factor Monoclonal Antibody vs Immune Checkpoint Inhibitors
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Tianxin Chen, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: KY2023-R206
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: AKI Incidence of Cancer Patients Receiving AntiVEGF or ICIs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AntiVEGF: cancer patients receiving anti-vascular endothelial growth factor monoclonal antibody (AntiVEGF)
  Interventions: Drug: AntiVEGF
- ICIs: cancer patients receiving immune checkpoint inhibitors (ICIs).
  Interventions: Drug: ICIs

INTERVENTIONS:
Drug: AntiVEGF — anti-vascular endothelial growth factor monoclonal antibody drug includes bevacizumab;
  Groups: AntiVEGF
Drug: ICIs — immune checkpoint inhibitors include Pembrolizumab, Sintilimab, toripalimab, Camrelizumab, Tislelizumab.
  Groups: ICIs

SUMMARY:
The goal of this a retrospective real-world study is to compare the AKI events in cancer patients receiving anti-vascular endothelial growth factor monoclonal antibody (AntiVEGF) vs immune checkpoint inhibitors (ICIs). The main question it aims to answer is whether the choice between AntiVEGF and ICIs affects the risks of acute kidney injury in cancer patients.

Cancer patients receiving AntiVEGF will be compared to those treated with ICIs to see if the AKI incidence is higher in patients receiving ICIs.

ELIGIBILITY:
Inclusion Criteria:

* Age >=20yr;
* Patients must have at least one "Evaluation and Management"visit with a diagnosis of cancer within 12 months before index date (In situ biopsy will not be required, since patients may receive a diagnosis from a biopsy of metastatic site);
* Indication to initiate AntiVEGF or ICIs

Exclusion Criteria:

* Patients without valid data and less than 3 months followup;
* Patients without baseline Scr value within 12 mon before index date;
* Patients with combination therapy of Anti-VEGF and ICIs ;
* Patients with chronic renal failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — >=20yr
Study Population: patients with malignancies treated with AntiVEGF or ICIs between Jan 2020 and December 2022
Sampling Method: Probability Sample
Enrollment: 1581 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
accumulative incidence of sustained AKI | 12 months after index date
  sustained AKI will be defined as the elevation ≥1.5 times baseline sCr for ≥72hours according to the Kidney Disease Improving Global Outcomes (KDIGO) sCr criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HR, Sugawara S, Lee JS, Kang JH, Inui N, Hida T, Lee KH, Yoshida T, Tanaka H, Yang CT, Nishio M, Ohe Y, Tamura T, Yamamoto N, Yu CJ, Akamatsu H, Takahashi S, Nakagawa K. First-line nivolumab, paclitaxel, carboplatin, and bevacizumab for advanced non-squamous non-small cell lung cancer: Updated survival analysis of the ONO-4538-52/TASUKI-52 randomized controlled trial. Cancer Med. 2023 Aug;12(16):17061-17067. doi: 10.1002/cam4.6348. Epub 2023 Aug 28. PMID 37641544
- [Background] Holloway RW, Thaker P, Mendivil AA, Ahmad S, Al-Niaimi AN, Barter J, Beck T, Chambers SK, Coleman RL, Crafton SM, Crane E, Ramez E, Ghamande S, Graybill W, Herzog T, Indermaur MD, John VS, Landrum L, Lim PC, Lucci JA, McHale M, Monk BJ, Moore KN, Morris R, O'Malley DM, Reid TJ, Richardson D, Rose PG, Scalici JM, Silasi DA, Tewari K, Wang EW. A phase III, multicenter, randomized study of olvimulogene nanivacirepvec followed by platinum-doublet chemotherapy and bevacizumab compared with platinum-doublet chemotherapy and bevacizumab in women with platinum-resistant/refractory ovarian cancer. Int J Gynecol Cancer. 2023 Sep 4;33(9):1458-1463. doi: 10.1136/ijgc-2023-004812. PMID 37666539
- [Background] Watanabe J, Muro K, Shitara K, Yamazaki K, Shiozawa M, Ohori H, Takashima A, Yokota M, Makiyama A, Akazawa N, Ojima H, Yuasa Y, Miwa K, Yasui H, Oki E, Sato T, Naitoh T, Komatsu Y, Kato T, Hihara M, Soeda J, Misumi T, Yamamoto K, Akagi K, Ochiai A, Uetake H, Tsuchihara K, Yoshino T. Panitumumab vs Bevacizumab Added to Standard First-line Chemotherapy and Overall Survival Among Patients With RAS Wild-type, Left-Sided Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA. 2023 Apr 18;329(15):1271-1282. doi: 10.1001/jama.2023.4428. PMID 37071094
- [Background] Bond MJG, Bolhuis K, Loosveld OJL, de Groot JWB, Droogendijk H, Helgason HH, Hendriks MP, Klaase JM, Kazemier G, Liem MSL, Rijken AM, Verhoef C, de Wilt JHW, de Jong KP, Gerhards MF, van Amerongen MJ, Engelbrecht MRW, van Lienden KP, Molenaar IQ, de Valk B, Haberkorn BCM, Kerver ED, Erdkamp F, van Alphen RJ, Mathijssen-van Stein D, Komurcu A, Lopez-Yurda M, Swijnenburg RJ, Punt CJA; Dutch Colorectal Cancer Study Group. First-line systemic treatment strategies in patients with initially unresectable colorectal cancer liver metastases (CAIRO5): an open-label, multicentre, randomised, controlled, phase 3 study from the Dutch Colorectal Cancer Group. Lancet Oncol. 2023 Jul;24(7):757-771. doi: 10.1016/S1470-2045(23)00219-X. Epub 2023 Jun 14. PMID 37329889
- [Background] Mantia CM, McDermott DF. Vascular endothelial growth factor and programmed death-1 pathway inhibitors in renal cell carcinoma. Cancer. 2019 Dec 1;125(23):4148-4157. doi: 10.1002/cncr.32361. Epub 2019 Sep 18. PMID 31532565
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Hanna RM, Barsoum M, Arman F, Selamet U, Hasnain H, Kurtz I. Nephrotoxicity induced by intravitreal vascular endothelial growth factor inhibitors: emerging evidence. Kidney Int. 2019 Sep;96(3):572-580. doi: 10.1016/j.kint.2019.02.042. Epub 2019 Apr 9. PMID 31229276
- [Background] Takada H, Yamashita K, Osawa L, Komiyama Y, Nakakuki N, Muraoka M, Suzuki Y, Sato M, Takano S, Fukasawa M, Yamaguchi T, Maekawa S, Takahashi K, Uchimura K, Enomoto N. Impact of Renal Function on the Prognosis of Patients Receiving Atezolizumab/Bevacizumab Combination Therapy and Lenvatinib Monotherapy for Unresectable Hepatocellular Carcinoma. Oncology. 2023;101(10):609-623. doi: 10.1159/000531111. Epub 2023 Jun 6. PMID 37279708
- [Background] Shye M, Hanna RM, Patel SS, Tram-Tran N, Hou J, Mccannel C, Khalid M, Hanna M, Abdelnour L, Kurtz I. Worsening proteinuria and renal function after intravitreal vascular endothelial growth factor blockade for diabetic proliferative retinopathy. Clin Kidney J. 2020 Jun 28;13(6):969-980. doi: 10.1093/ckj/sfaa049. eCollection 2020 Dec. PMID 33391740
- [Derived] Zhu J, Ding X, Zhang J, Chen B, You X, Chen X, Chen T. Acute kidney injury in cancer patients receiving anti-vascular endothelial growth factor monoclonal antibody vs. immune checkpoint inhibitors: a retrospective real-world study. BMC Cancer. 2024 Jun 24;24(1):756. doi: 10.1186/s12885-024-12540-y. PMID 38914959